CLINICAL TRIAL: NCT01273428
Title: Comparison of HP011-101, HP828-101, and Standard Care in the Management of Stage I-II Pressure Ulcers in Patients With Spinal Cord Injury
Brief Title: HP011-101, HP828-101, and Standard Care for Pressure Ulcers
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: The device test article is no longer available
Sponsor: Healthpoint (Industry)
Responsible Party: Herbert B. Slade, MD FAAAAI / Chief Medical Officer, Healthpoint, Ltd
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 011-101-09-041
Record Dates: First submitted 2010-12-03; First posted 2011-01-10 (Estimated); Last update posted 2012-09-12 (Estimated); Status verified 2011-01

CONDITIONS: Pressure Ulcers
MeSH Terms: conditions — Pressure Ulcer | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- HP011-101 (Active Comparator)
  Interventions: Drug: HP011-101
- HP828-101 (Active Comparator)
  Interventions: Device: HP-828-101
- Standard Care (Other)
  Interventions: Other: Standard Care

INTERVENTIONS:
Drug: HP011-101
  Arms: HP011-101
Device: HP-828-101
  Arms: HP828-101
Other: Standard Care
  Arms: Standard Care

SUMMARY:
Testing a drug and a device for the treatment of pressure ulcers, compared with current treatments.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must meet all of the following criteria to be eligible for the study:
* Provide informed consent, or informed assent if less than 18 years of age.
* Age 12 years or older, of either sex, and of any race or skin type, provided that their skin color, in the opinion of the Investigator, will not interfere with the study assessments.
* Have a pressure ulcer ≥ 5 cm² and ≤ 100 cm² in area (measured as greatest length x perpendicular width of the area of non-blanching erythema or denuded skin, whichever is greater), and will remain hospitalized for at least three weeks.
* Are capable of maintaining an adequate nutritional status.
* All female subjects must have a negative urinary pregnancy test.
* Have, within 12 weeks prior to screening, clinical laboratory test results indicating:

  * Serum albumin ≥ 3.0 g/dL (30 g/L)
  * Alkaline phosphatase, ALT, AST, BUN and serum creatinine levels < 3x upper limit of the Healthpoint normal range (refer to Section 18.1.2)
  * HbA1C ≤ 12%
  * Hemoglobin ≥ 10 g/dL
* The most recently obtained values must be evaluated against these criteria. If these values are not available from a blood sample within 12 weeks of screening, blood must be drawn at screening and these laboratory values determined.
* For ulcers that will require surgical debridement prior to enrollment, the wound must be expected to remain a Stage I or Stage II partial thickness wound after debridement.

Exclusion Criteria:

* Subjects meeting any of the following criteria are not eligible to enter the study:
* Have a known hypersensitivity to any of the test articles or their components.
* Have received therapy with another investigational agent within thirty (30) days of screening.
* Are pregnant or nursing.
* Are currently being treated with systemic antibiotics.
* Have received systemic treatment with glucocorticoids for > 10 consecutive days within 1 month prior to the start of the study.
* Have received chemotherapy or radiation therapy within the past 5 years.
* Have clinical evidence of bacterial or fungal infection of the wound per visual/clinical assessment.
* Have a severe burn, immunodeficiency disorder, hematologic disorder, or metastatic malignancy.
* Have had documented osteomyelitis in the wound area within 6 months prior to screening.
* The Principal Investigator may declare any subject ineligible for a valid medical reason.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Primary Completion 2011-06 (Estimated); Study Completion 2011-11 (Estimated)

PRIMARY OUTCOMES:
Change in Wound Bed Scores | 22 days

SECONDARY OUTCOMES:
Adverse Events | 22 days

CONTACTS AND LOCATIONS:
Overall Officials: Herbert B Slade, MD, Study Chair — Healthpoint, Ltd